CLINICAL TRIAL: NCT03957603
Title: Effects of Medical Nutrition Therapy Combined With TPF-DM in Pregnant Women With Gestational Diabetes Mellitus on Blood Glucose Fluctuations and Pregnancy Outcomes
Brief Title: Medical Nutrition Therapy Combined With TPF-DM in Pregnant Women With Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Zhejiang University School of Medicine, Obstetrics and Gynecology Hospital (Unknown); Nutricia Pharmaceutical Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Guanghui Li, Professor, MD, PhD, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-KY-061-01
Record Dates: First submitted 2019-05-14; First posted 2019-05-21 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Medical Nutrition Therapy; Gestational Diabetes Mellitus; Adverse Pregnancy Outcomes; Fasting Plasma Glucose; HbA1c; Gestational Weight Gain
MeSH Terms: conditions — Diabetes, Gestational; Gestational Weight Gain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPF-DM Combined with Medical Nutrition Therapy Intervention (Experimental): Participants in the experimental group will be provided with an individualized dietary, nutrition recommendation and the additional Enteral Nutrition Suspension (TFP-DM, Diason 0.75 kcal/ml). Participants are required to schedule the first follow-up visit one week after receiving the individualized recommendations. Afterward, the regularly scheduled follow-up visit will be scheduled every two to four weeks.
  Interventions: Dietary Supplement: Enteral Nutrition Suspension (TFP-DM)
- Medical Nutrition Therapy Intervention (Active Comparator): Based on the standard care, Participants will receive an individualized dietary, nutrition recommendations with the application of food exchange porting. Participants are required to schedule the first follow-up visit one week after receiving the individualized recommendations. Afterward, the regularly scheduled follow-up visit will be scheduled every two to four weeks.
  Interventions: Behavioral: Medical Nutrition Therpay

INTERVENTIONS:
Dietary Supplement: Enteral Nutrition Suspension (TFP-DM) — Individualized dietary and lifestyle intervention combined with the recommendation of Enteral Nutrition Suspension (TPF-DM, Diason 0.75 kcal/ml)
  Arms: TPF-DM Combined with Medical Nutrition Therapy Intervention
Behavioral: Medical Nutrition Therpay — Individualized dietary and lifestyle intervention
  Arms: Medical Nutrition Therapy Intervention

SUMMARY:
Background:

Gestational diabetes mellitus (GDM), GDM is the first time of gestational impaired glucose tolerance in pregnant women. It is the most common complication disease in women of childbearing age. It is associated with the high risk of adverse health outcomes for both mothers and offsprings and the variety of metabolic disease, including type 2 diabetes, etc. As for the epidemiology data of GDM in China, the prevalence is around 18% based on the criteria from the International Association of Diabetes in Pregnancy Study Groups, IADPSG. Several studies claimed that the diabetes-specific formula improved glycemic control in type 2 diabetes patients. However, the effects of medical nutrition therapy combined with the diabetes-specific formula in pregnant women with gestational diabetes mellitus (GDM) are unclear.

Objective:

This study examines whether medical nutrition therapy combined with Enteral Nutrition Suspension (TFP-DM, Diason 0.75 kcal/ml) in GDM women could improve the glycemic control and the pregnancy outcomes.

DETAILED DESCRIPTION:
Design:

A randomized controlled trial in pregnant women with gestational diabetes mellitus (GDM) will be performed at 24-28 weeks of gestation until the 42 days after delivery. Participants will be randomly assigned to the control group (Medical Nutrition Therapy) or the intervention group (Medical Nutrition Therapy combined with TFP-DM). The control group will receive the individualized Medical Nutrition Therapy, which focuses on restricting energy intake combined with behavioral lifestyle modification through participation in group sessions and individual counseling. The intervention group has two components. The first part has the same intervention with the control group. The second part has the additional Enteral Nutrition Suspension (TFP-DM, Diason 0.75 kcal/ml) intervention based on the standard Medical Nutrition Therapy. It meant 200ml/150Kcal TFP-DM will be suggested to participants in the intervention group 2 times per day. The 400ml TFP-DM will replace the 25 grams of grains and dairies during breakfast and the snack session after dinner. Overall, the control group and the intervention group will receive the same amount of carbohydrate and calorie intake. The primary outcome will be fasting plasma glucose concentration, HbA1c concentration. The secondary outcome will be serum glycated albumin, serum insulin concentration, the rate of using insulin for patients, the insulin sensitivity (HOMA-IS), the gestational weight gain, the incidence of macrosomic infants.

Hypothesis:

Medical nutrition therapy combined with the enteral nutrition suspension (TFP-DM, Diason 0.75 kcal/ml) in pregnant women with gestational diabetes mellitus (GDM) will improve in glucose and lipid metabolism and the relevant adverse pregnancy outcomes, and provide the evidence-based in clinical nutrition therapy for gestational diabetes mellitus (GDM) disease.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 24 and 28 weeks of gestation
* Age >= 18 years
* Singleton pregnancy
* Two of three or three results of the oral glucose tolerance test (OGTT) are above the diagnostic criteria. (The diagnostic criteria for three results of OGTT: Fasting plasma glucose ≥ 5.1mmol/L, 1-hour OGTT plasma glucose ≥ 10.0mmol/L, 2-hour OGTT plasma glucose ≥ 8.5mmol/L)

Exclusion Criteria:

* History of prenatal hypertension, diabetes, hyperlipidemias, liver disease, kidney disease, digestive tract disease and infectious disease (hepatitis, tuberculosis etc.)
* Gestational weeks < 24 or > 28
* Age < 18 years or Age > 45 years
* Multiple pregnancy
* Food allergic history
* Regular smoking, drinking alcohol
* Patients with the history of using the assisted reproductive technology
* Patients with psychiatric disorders that prevents correctly answer the questions
* Patients who are unable to answer the questionnaire questions
* Bariatric surgery history
* Non-adherence of dietary and lifestyle recommendation
* Threatened abortion

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from Baseline at 2 months | Gestational age 24-28 weeks and 32-34 weeks and 36-40 weeks and 42-70 days after delivery
Insulin treatmeant ratio | From enrollment to delivery
Change in serum glycated albumin from Baseline at 2 months | Gestational age 24-28weeks and 32-34weeks and 36-40 weeks and 42-70days after delivery
Change in fasting blood glucose concentration from Baseline at 2 months | Gestational age 24-28 weeks and 32-34 weeks and 36-40 weeks and 42-70 days after delivery
Change in Fasting insulin concentration from Baseline at 2 months | Gestational age 24-28 weeks and 32-34 weeks and 36-40 weeks and 42-70 days after delivery

SECONDARY OUTCOMES:
Oral glucose tolerance test | Gestational age 24-28 weeks and 42-70 days after delivery
The insulin sensitivity (HOMA-IS) | From enrollment to the 42 days after delivery
Gestational weight gain | From enrollment to the 42 days after delivery
The incidence of macrosomia infants | From enrollment to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Guanghui Li, MD, PhD, Principal Investigator — Beijing Obstetrics and Gynecology Hospital
Locations (1):
- Beijing Obstetrics and Gynecology Hospital,Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Yang R, Han W, Zheng W, Xu D, He J, Yuan X, Zhang L, Tian Z, Li G. Administration of a diabetes-specific formula can improve postprandial glycemic control and delay insulin use in gestational diabetes mellitus: A randomized controlled trial from two centers. Clin Nutr. 2024 Dec;43(12):265-274. doi: 10.1016/j.clnu.2024.11.001. Epub 2024 Nov 6. PMID 39536397